CLINICAL TRIAL: NCT04403789
Title: Effects of a Workplace Exercise Intervention on Cardio-Metabolic Health: Randomized Controlled Trial
Brief Title: Effects of a Workplace Exercise Intervention on Cardio-Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Collaborators: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Javaid Nauman, Assistant Professor, United Arab Emirates University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23081010
Record Dates: First submitted 2020-05-06; First posted 2020-05-27 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Risk Factor; Pre Diabetes; High Blood Pressure; Elevated LDL Cholesterol
Keywords: cardiometabolic risk factors and exercise; workplace intervention
MeSH Terms: conditions — Glucose Intolerance; Hypertension; Hyperlipoproteinemia Type II; Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention The intervention duration is 12 weeks and it will provide the employees exercise time of 2 hours per week. The 2 hours should be used in two days either at the middle or at the end of working hours. The 2-hours exercise session will be conducted under the supervision of a certified trainer in the gym workplace. The 12 weeks period was chosen based on recommendations from previous studies to examine the effect of exercise interventions. The delayed intervention group will be asked to perform their usual routine and continue their usual exercise/physical activity routines. However, after the intervention is completed the delayed intervention group will also receive 2 hours of exercise time per week from working hours for 4 weeks. The reason for this is to encourage participants to participate in the study regardless of which group they will be assigned in. Also, this will help us reduce contamination as participants will not be aware which group they were assigned in.
Who Masked: Participant
Masking Description: Single blinding was used. The intervention group was renamed Group A and the delayed-intervention group as Group B to blind participants from the intervention. Participants were strongly encouraged not to disclose their allocation status during the health measurement assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): During the intervention period they will receive 2 hours per week of group exercise sessions during working hours for 12 weeks. However, after the intervention period, there will be no change in working hours
  Interventions: Other: Exercise Time; Behavioral: Supervised Group Exercise
- Delayed Intervention Group (Control group) (Active Comparator): During the intervention period there will be no change in working hours. However, after the intervention period they will receive 2 hours of exercise time during working hours per week for 4 weeks
  Interventions: Other: Exercise Time

INTERVENTIONS:
Other: Exercise Time — Employees will be provided with exercise time of 2 hours per week. The 2 hours should be used in two days. The intervention duration is 12 weeks.
  Other Names: Working hours
Behavioral: Supervised Group Exercise — The intervention group will receive 2-hours of exercise sessions per week under the supervision of a certified trainer in the gym workplace. The intervention duration is 12 weeks.
  Other Names: Group exercise sessions
  Arms: Intervention Group

SUMMARY:
Background: The rising levels of physical inactivity in the Eastern Mediterranean region (43.2%) and in the United Arab Emirates (38%) compared with the global levels of physical inactivity (31.2%) is alarming (6,15). Therefore, action is required to reduce physical inactivity using evidence-based strategies. This study aims to provide scientific evidence that if the workplace environment promotes behavior change, physical activity levels could increase and, therefore, improve health. Objective: Primary objective: to determine whether the workplace exercise intervention will improve the cardio-metabolic risk components for the employees. Secondary objective: to determine whether the workplace exercise intervention will improve physical activity levels even after 4 weeks of completing the intervention. Methods: A total of 150 participants will be recruited from a semi-government telecommunication company after meeting the eligibility criteria; 75 will be assigned to the intervention group and 75 to the delayed intervention group. Intervention: The Intervention group will receive 2 hours of exercise per week during working hours for 12 weeks. One hour can be used per day. The intervention group will be assigned to attend personal trainer sessions in the workplace gym during the intervention. After the intervention is completed the delayed intervention group will also receive 2 hours of exercise time per week from working hours for 4 weeks. Expected results: There is a statistically significant difference in the primary and secondary health outcome between the intervention group and delayed intervention group. Expected conclusion: Increasing exercise time in the workplace is associated with favorable cardio-metabolic risk profile.

DETAILED DESCRIPTION:
Study Design The study is considered a parallel randomized controlled trial with a 1:1 allocation ratio to intervention group and delayed intervention group.

Recruitment An invitation to attend an informational session will be sent to the employees in the company's headquarter building in Dubai, United Arab Emirates. The invitation will emphasize that participation is voluntary and that participants can withdraw at any time without giving any reason. The informational session will discuss the study details (e.g. eligibility criteria) and some tips for physical activity. All employees who wish to participate will need to sign a consent form. The participants who are eligible will have to take an appointment in the workplace health center to make the required health measurements. A total of 150 participants will be recruited for the study. The eligibility of joining the workplace intervention will be based on the eligibility criteria listed below.

Setting and location The intervention will be conducted in the headquarter building of a semi-government telecommunication company in Dubai, United Arab Emirates. The headquarter building includes a gym and swimming pool. The intervention will use the gym workplace for conducting the exercise sessions.

Sample Size Previous studies concerning physical activity and cardiometabolic risk factors used 80% to 91% power and effect sizes ranging between 0.51 and 1.82 to find a significant difference between groups (8,10, 12-13). There are various reasons for choosing these articles for sample size calculations. For example, one article used a 12-week physical activity intervention and offered 3 sessions of physical activity per week (13). The same article included healthy adult participants (13). In addition, the cited articles were concerned with the effect of exercise on specific metabolic risk factors. These metabolic risk factors were waist circumference, systolic blood pressure. fasting glucose, lipid profiles (8,10, 12-13). More specifically, one article focused on waist circumference and physical activity (8). In contrast another article focused on systolic blood pressure and physical activity (10). For the present study, 124 participants will be required at 80% power. A further 20% more participants will be added because it is expected that participants might drop out during the intervention. Therefore, the investigators will recruit a total of 150 participants. The intervention group will have 75 participants and the delayed intervention group will have 75 participants.

Statistical Analysis Analyses and reporting will be in line with CONSORT guidelines, with all analyses being on an intention-to-treat principle regardless of intervention compliance. For a comparison between intervention and delayed intervention arms of the 12- weeks change in outcomes, the investigators plan to use analysis of covariance model, with baseline values as the covariate to control for chance imbalances at baseline. Age and sex specific interaction analyses will be conducted. In addition, the investigators will adopt a linear mixed model approach to provide the mean intervention effect, and quantification of individual differences in response to the intervention. The clinical significance of the intervention effect will be elaborated with magnitude-based inferences, confidence intervals, and confidence levels. Accepted regression modelling methods will be used to explore the intervention effects on the secondary objectives. Multiple imputation techniques will assess the sensitivity of the analyses to the missing at random assumption. Significance tests at 5%, either t-test or chi squared tests will be used to compare those with complete data and those who have missing outcomes. Finally, the investigators will develop a detailed coding scheme and coding checking protocol, cross tabulation, negative case analysis and respondent validation to enhance dependability and trustworthiness.

Evaluation

The completion of the tasks in the study will evaluate its success. For example:

Inviting all employees to the informational session and selecting eligible participants.

Randomly allocating participants to the intervention and delayed intervention group Collecting and analyzing blood samples pre and post the intervention period. Physical activity levels recorded through IPAQ and accelerometer. Recording participants attendance to personal trainer sessions. The evaluation of the intervention program will also depend on the primary and secondary health outcomes of the participants in the intervention and delayed intervention group. If there is a significant difference between the health outcomes of the two groups then the workplace intervention would have a positive effect.

Data Management The study investigators will ensure that the participants' anonymity is maintained. All data will be stored securely in an electronic database. Participants will be assigned a unique research number on the electronic database. No individually identifiable information will be included in the research database. The research number link to personal identifying information will be maintained in a secure server physically separate from the electronic database, which will be accessible only by specifically designated staff. This secure linkage will allow for the subsequent addition of new information to the research database, while maintaining no personal identifiers in the research database. Questionnaire responses and physical measures will be maintained under the unique research number.

Informed Consent The participant must personally sign and date (on paper or electronically) the latest approved version of the Informed Consent form before any study specific procedures are performed. Written versions of the Participant Information Leaflet and Informed Consent will be presented to the participants detailing no less than: the exact nature of the study; what it will involve for the participant; the implications and constraints of the protocol; the known side effects and any risks involved in taking part. It will be clearly stated that the participant is free to withdraw from the study at any time for any reason without prejudice to future care, and with no obligation to give the reason for withdrawal. The participant will be allowed as much time as wished to consider the information, and the opportunity to question the investigator or other independent parties to decide whether the participant will enroll in the study. Written Informed Consent will then be obtained by means of participant-dated signature and dated signature of the person who presented and obtained the Informed Consent. The person who obtained the consent must be suitably qualified and experienced, and have been authorized to do so by the Principal Investigator. A copy of the signed Informed Consent will be given to the participant.

Patient confidentiality and data security Patient names and identifying numbers (medical record number, Emirates Identification Card number etc.) will be removed from each record and replaced by a unique study number. It will not be possible for the researchers to identify the patients. Data will be held on the hard-drive of the researcher's computer in a locked office.

Discontinuation/Withdrawal of Participants from Study Each participant has the right to withdraw from the study at any time without giving any reason. Should a participant wish to withdraw from the study, they are advised in the participant information leaflet to contact the study coordinator. Should the participant wish for xx samples and data collected to be destroyed this will be done in a prompt and secure manner and a message will be sent to the person to confirm this. The reason for withdrawal, if given, will be recorded in the database.

Expenses and Benefits There is no plan to offer any monetary compensation to participants but if recruitment rates are lower than required, the investigators will pilot whether offering free (non-monetary) gifts, certificates, first aid kits, etc. improves response rates or not. For example, there will be one week where there are no gifts and another week where gifts are provided and see how that affects response rates.

Risks and Benefits Assessment The main risks of participation are direct physical harm and breaches of privacy/confidentiality. The risks of direct physical harm are minimal. All clinical staff will receive full training on all of the study procedures, and all measurements will be performed by trained staff/nurses. The exercise session will be conducted under supervision of certified personal trainers to ensure proper exercise techniques and therefore reduce risk of any potential injury. Participant's health information will be protected by restricted access and through use of de-identified labelling and use of de-identified data sets for analysis.

There are direct benefits to the individuals involved, together with the satisfaction of contributing to societal benefit by the increased understanding of role of exercise at workplace to improve health. The benefits of this study for science and society include but not limited to increase the investigators knowledge of the role of physical activity on overall health status, and risk factors for cardiovascular disease. The study aims to provide direction for prevention programs, particularly in the office workers/employees who are the key target group for interventions aiming to identify long lasting ways to increase participation in physical activity with potential health benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be an employee in the company and have at least a waist circumference of ≥94 cm (≥90 cm for South and East Asians) for males and ≥ 80 cm for females.
2. Aged 18 to 59 years old.
3. Availability of the participants for the study duration.
4. Participant is willing to commit to the intervention until the end.
5. Signed written consent to participate.

Exclusion Criteria:

1. Severe injury in the joints or the back or any medical condition that would prevent them from exercising, or the participant is advised not to exercise by a doctor.
2. Pregnant.
3. Any planned major surgical procedures during the intervention period.
4. Self-reported cardiovascular disease, lung disease, or cancer.
5. Currently participating in a health promotion program

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline high Blood Pressure (mmHg) at 12 Weeks | The outcome will be measured for both groups at baseline and after the 12-week intervention.
  Primary objective: to determine whether the workplace exercise intervention will improve the cardio-metabolic risk components for the employees. The cardio-metabolic risk components compromises of several risk factors including, high blood pressure.
  Measurement Criteria:
  Systolic blood pressure ≥ 130 mm Hg OR Diastolic blood pressure ≥ 85 mm Hg
Change from Baseline Waist Circumference (centimetres) at 12 Weeks | The outcome will be measured for both groups at baseline and after the 12-week intervention.
  Primary objective: to determine whether the workplace exercise intervention will improve the cardio-metabolic risk components for the employees. The cardio-metabolic risk components compromises of several risk factors including, waist circumference above normal range. The waist circumference criteria are:
  Measurement Criteria:
  1-Waist circumference above normal (cm): > 102 cm for males and > 88 cm for females (9)
Change from Baseline HDL-cholesterol (mmol/L) at 12 Weeks | The outcome will be measured for both groups at baseline and after the 12-week intervention.
  Primary objective: to determine whether the workplace exercise intervention will improve the cardio-metabolic risk components for the employees. The cardio-metabolic risk components compromises of several risk factors including, elevated HDL-cholesterol.
  Measurement Criteria:
  < 40 mg/dL in males and < 50 mg/dL in females.
Change from Baseline Triglycerides (mg/dL) at 12 Weeks | The outcome will be measured for both groups at baseline and after the 12-week intervention.
  Primary objective: to determine whether the workplace exercise intervention will improve the cardio-metabolic risk components for the employees. The cardio-metabolic risk components compromises of several risk factors including, Elevated Triglycerides (mg/dL)
  Measurement Criteria:
  • Elevated Triglycerides ≥ 150 (mg/dL)
Change from Baseline Fasting Plasma Glucose (mmol/L) at 12 Weeks | The outcome will be measured for both groups at baseline and after the 12-week intervention.
  Primary objective: to determine whether the workplace exercise intervention will improve the cardio-metabolic risk components for the employees. The cardio-metabolic risk components compromises of several risk factors including, pre-diabetes (Fasting plasma glucose).
  Measurement Criteria:
  1-Pre-diabetes: Fasting plasma glucose (mg/dL) ≥ 100 mg/dL

SECONDARY OUTCOMES:
Change from Baseline Physical Activity (IPAQ Questionnaire) at 12 Weeks and 16 weeks | This outcome will be measured for both groups at baseline, at 12-week intervention. The third measurement will be at 16 weeks (4 weeks after completing the intervention, for the intervention group only).
  Secondary objective:To determine whether the workplace exercise intervention will improve physical activity levels after 4 weeks of completing the intervention. Two measurement criteria will be used to measure physical activity in this study. One of these measurements is the International Physical Activity Questionnaire (IPAQ). This measurement classifies participants into three categories based on the answers provided:
  1. Low physical activity
  2. Moderate physical activity
  3. High physical activity (7)
Change from Baseline Physical Activity (AX3 Device) at 12 Weeks and 16 weeks | This outcome will be measured for both groups at baseline, at 12-week intervention. The third measurement will be at 16 weeks (4 weeks after completing the intervention, for the intervention group only).
  Secondary objective: To determine whether the workplace exercise intervention will improve physical activity levels after 4 weeks of completing the intervention. Two measurement criteria will be used to measure physical activity in this study. One of these measurements is the AX3 (3-Axis Logging Accelerometer). The accelerometer devices will be configured to capture three-dimensional acceleration at 100 Hz with a dynamic range of ±8 g.

CONTACTS AND LOCATIONS:
Overall Officials: Javaid Nauman, PhD, Principal Investigator — United Arab Emirates University
Locations (1):
- Emirates Integrated Telecommunication Company (Du), Headquarters Building., Dubai, Dubai Internet City, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to publish the study protocol. The data will be available if approval from Dubai Scientific Research Ethics Committee in Dubai Health Authority is acquired.
Supporting Information: Study Protocol
Time Frame: Data availability begins one year after publication. Data availability ends three years after publications
Access Criteria: To researchers who provide a methodologically sound proposal and has approval from Dubai Scientific Research Ethics Committee in Dubai Health Authority.

REFERENCES:
- [Background] Axivity Ltd. AX3 [Internet]. AX3. 2019 [cited 2019 Jun 16]. Available from: http://www.axivity.com/product/1
- [Background] Bergman F, Wahlstrom V, Stomby A, Otten J, Lanthen E, Renklint R, Waling M, Sorlin A, Boraxbekk CJ, Wennberg P, Ohberg F, Levine JA, Olsson T. Treadmill workstations in office workers who are overweight or obese: a randomised controlled trial. Lancet Public Health. 2018 Nov;3(11):e523-e535. doi: 10.1016/S2468-2667(18)30163-4. Epub 2018 Oct 12. PMID 30322782
- [Background] Cannon CP. Cardiovascular disease and modifiable cardiometabolic risk factors. Clin Cornerstone. 2007;8(3):11-28. doi: 10.1016/s1098-3597(07)80025-1. PMID 18452839
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1046-e1081. doi: 10.1161/CIR.0000000000000624. Epub 2018 Nov 10. No abstract available. PMID 30565953
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Worldwide trends in insufficient physical activity from 2001 to 2016: a pooled analysis of 358 population-based surveys with 1.9 million participants. Lancet Glob Health. 2018 Oct;6(10):e1077-e1086. doi: 10.1016/S2214-109X(18)30357-7. Epub 2018 Sep 4. PMID 30193830
- [Background] International Physical Activity Questionnaire. IPAQ scoring protocol - International Physical Activity Questionnaire [Internet]. 2005 [cited 2019 Jan 27]. Available from: https://sites.google.com/site/theipaq/scoring-protocol
- [Background] Irving BA, Davis CK, Brock DW, Weltman JY, Swift D, Barrett EJ, Gaesser GA, Weltman A. Effect of exercise training intensity on abdominal visceral fat and body composition. Med Sci Sports Exerc. 2008 Nov;40(11):1863-72. doi: 10.1249/MSS.0b013e3181801d40. PMID 18845966
- [Background] Klein S, Allison DB, Heymsfield SB, Kelley DE, Leibel RL, Nonas C, Kahn R; Association for Weight Management and Obesity Prevention; NAASO; Obesity Society; American Society for Nutrition; American Diabetes Association. Waist circumference and cardiometabolic risk: a consensus statement from shaping America's health: Association for Weight Management and Obesity Prevention; NAASO, the Obesity Society; the American Society for Nutrition; and the American Diabetes Association. Diabetes Care. 2007 Jun;30(6):1647-52. doi: 10.2337/dc07-9921. Epub 2007 Mar 14. No abstract available. PMID 17360974
- [Background] Molmen-Hansen HE, Stolen T, Tjonna AE, Aamot IL, Ekeberg IS, Tyldum GA, Wisloff U, Ingul CB, Stoylen A. Aerobic interval training reduces blood pressure and improves myocardial function in hypertensive patients. Eur J Prev Cardiol. 2012 Apr;19(2):151-60. doi: 10.1177/1741826711400512. Epub 2011 Mar 4. PMID 21450580
- [Background] Nichols GA, Horberg M, Koebnick C, Young DR, Waitzfelder B, Sherwood NE, Daley MF, Ferrara A. Cardiometabolic Risk Factors Among 1.3 Million Adults With Overweight or Obesity, but Not Diabetes, in 10 Geographically Diverse Regions of the United States, 2012-2013. Prev Chronic Dis. 2017 Mar 9;14:E22. doi: 10.5888/pcd14.160438. PMID 28278130
- [Background] Tomeleri CM, Ribeiro AS, Souza MF, Schiavoni D, Schoenfeld BJ, Venturini D, Barbosa DS, Landucci K, Sardinha LB, Cyrino ES. Resistance training improves inflammatory level, lipid and glycemic profiles in obese older women: A randomized controlled trial. Exp Gerontol. 2016 Nov;84:80-87. doi: 10.1016/j.exger.2016.09.005. Epub 2016 Sep 9. PMID 27616162
- [Background] Tomeleri CM, Souza MF, Burini RC, Cavaglieri CR, Ribeiro AS, Antunes M, Nunes JP, Venturini D, Barbosa DS, Sardinha LB, Cyrino ES. Resistance training reduces metabolic syndrome and inflammatory markers in older women: A randomized controlled trial. J Diabetes. 2018 Apr;10(4):328-337. doi: 10.1111/1753-0407.12614. Epub 2017 Dec 11. PMID 29031002
- [Background] WHO. WHO | Waist circumference and waist-hip ratio [Internet]. WHO. 2008 [cited 2018 Dec 12]. Available from: http://www.who.int/nutrition/publications/obesity/WHO_report_waistcircumference_and_waisthip_ratio/en/
- [Background] WHO. United Arab Emirates health profile 2015 [Internet]. 2016. Available from: http://applications.emro.who.int/dsaf/EMROPUB_2016_EN_19276.pdf
- [Derived] Alrahma AM, Habib MA, Oulhaj A, Loney T, Boillat T, Shah SM, Ahmed LA, Nauman J. Effects of a workplace exercise intervention on cardiometabolic health: study protocol for a randomised controlled trial. BMJ Open. 2021 Nov 3;11(11):e051070. doi: 10.1136/bmjopen-2021-051070. PMID 34732483